CLINICAL TRIAL: NCT04748393
Title: Risk, Predictors, Impact and Outcome of Anticoagulation-associated Abnormal Menstrual Bleeding in Female Patients With VTE
Brief Title: Risk, Predictors, Impact and Outcome of Anticoagulation-associated Abnormal Menstrual Bleeding
Acronym: TEAM-VTE
Status: Terminated | Type: Observational
Why Stopped: Low enrolment
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Erik Klok, principal investigator, Leiden University Medical Center
Other Study IDs: LUMC2017132
Record Dates: First submitted 2019-08-14; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Venous Thromboembolism
Keywords: menorrhagia; anticoagulation
MeSH Terms: conditions — Venous Thromboembolism; Menorrhagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: Consecutive female patients between the ages of 18 and 50 with child bearing potential and objectivated, symptomatic VTE, who fulfil all the inclusion criteria and meet none of the exclusion criteria, are eligible for inclusion.

SUMMARY:
This study is an international, multicenter, academically sponsored, observational study, that focusses on fertile female patients with proven symptomatic deep vein thrombosis of the legs (DVT) or acute pulmonary embolism (PE). The incidence and severity of abnormal menstrual bleeding will be assessed for each menstrual period and correlated to quality of life. Causes of abnormal menstrual bleeding other than active anticoagulant treatment will be assessed. Treatment of abnormal menstrual bleeding (all within routine clinical care) will be evaluated for efficacy and safety.

DETAILED DESCRIPTION:
A recently performed international survey of expert opinion and current practice revealed divergent expert recommendations and very heterogeneous management approach in clinical practice with regard to anticoagulation choice, use of HC and treatment of abnormal uterine bleeding during anticoagulant treatment of VTE. Together with the fact that up to 70% of female patients with childbearing potential treated with anticoagulants may suffer from abnormal menstrual bleeding with a severe negative impact on quality of life, this is a compelling argument to initiate high quality observational studies to better quantify the magnitude of the problem and to identify unmet clinical needs. This study will do so and at the same time provide solid ground for future prospective management trials aimed at establishing preventive and/or treatment strategies for VTE patients with anticoagulant-associated abnormal menstrual bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of subject to understand the character and individual consequences of this clinical study;
2. Signed and dated informed consent of the subject available before the start of any specific study procedures;
3. Age ≥18 years and ≤ 50 years;
4. Confirmed symptomatic first or recurrent VTE;

   1. DVT: incompressibility of proximal or distal veins of the affected leg by compression ultrasonography or venous filling defect on multi-detector computed tomography venography. The diagnosis of ipsilateral recurrent DVT is defined as a CUS that shows incompressibility of a different venous segment than at the reference CUS examination, or in case of a pronounced increase in vein diameter (≥4 mm) of a previous non-compressible venous segment, or by an abnormal signal of Magnetic resonance direct thrombus imaging (MRDTI);
   2. PE: both first and recurrent PE are diagnosed in case of at least one filling defect in the pulmonary artery tree on multi-detector computed tomography pulmonary angiography (CTPA) up to the subsegmental level, or high probability result of ventilation perfusion scintigraphy;
5. Childbearing potential, i.e. with active menstrual cycle with or without hormonal regulation of any kind initiated for reasons of either contraception or for treatment of abnormal menstrual bleeding;
6. Inclusion before the first day of next menstrual cycle after VTE diagnosis or within 1 month after the VTE diagnosis, whichever comes first.

Exclusion Criteria:

1. Woman between the ages of 18 and 50 who were subjected to hysterectomy or chemically induced menopause;
2. Woman between the ages of 18 and 50 with premature menopause (established before study inclusion);
3. Planned treatment with parenteral anticoagulation (and no switch to oral drugs);
4. Medical or psychological condition that would not permit completion of the study or signing of informed consent, including life expectancy less than 6 months, or unwillingness to sign informed consent;
5. Non-compliance or inability to adhere to the follow-up visits;
6. Pregnancy or post-partum (first three months) associated VTE;
7. Active in vitro fertilization (IVF) treatment or planned IVF treatment during the study period.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — female patients within their fertile age, diagnosed with acute venous thromboembolism
Study Population: Consecutive female patients between the ages of 18 and 50 with child bearing potential and objectivated, symptomatic VTE, who fulfil all the inclusion criteria and meet none of the exclusion criteria, are eligible for inclusion.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Primary objective | 3-month follow-up
  Rate of new-onset abnormal menstrual bleeding (PBAC >100 ml), and its impact on quality of life

CONTACTS AND LOCATIONS:
Overall Officials: F.A. Klok, Principal Investigator — LUMC Leiden
Locations (7):
- Medical University Hospital, Vienna, Austria
- France (2):
  - Hôpital de la Cavale Blanche, Brest
  - CHU Saint-Etienne, Saint-Etienne
- University Medical Centre Mannheim, Mannheim, Germany
- Leiden University Medical Center, Leiden, Netherlands
- Geneva University Hospital, Geneva, Switzerland
- Guy's & St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Derived] de Jong CMM, Blondon M, Ay C, Buchmuller A, Beyer-Westendorf J, Biechele J, Bertoletti L, Colombo G, Donadini MP, Hendriks SV, Jara-Palomares L, Nopp S, Ruiz-Artacho P, Stephan P, Tromeur C, Vanassche T, Westerweel PE, Klok FA. Incidence and impact of anticoagulation-associated abnormal menstrual bleeding in women after venous thromboembolism. Blood. 2022 Oct 20;140(16):1764-1773. doi: 10.1182/blood.2022017101. PMID 35925686